CLINICAL TRIAL: NCT05540444
Title: RadConnect Communication Application
Acronym: RadConnect
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000556
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Communication
Keywords: Radiologists; Radiology Technologists
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RadConnect — The study will be performed in a clinical setting at the department of radiology of LUMC, meaning that we aim to test the hypothesis that ("RadConnect") can reduce the number of phone calls from a select set of extension used by technologists (the "Sending Extensions") to another select set of extensions manned by radiologists ("Receiving Extensions").

SUMMARY:
The aim is to evaluate the impact of an innovative asynchronous communication application on the number of calls from technologists to radiologists. Even though it is paramount that radiologists be accessible and available to other healthcare workers in the enterprise, frequent interruptions have negative impact on productivity and well-being. A novel communication app was developed that streamlines communication between technologists and radiologists: RadConnect.

ELIGIBILITY:
Inclusion Criteria:

* Individuals that are employed by LUMC
* Individuals that are radiologists, radiology fellows, radiology residents, radiology technologists, doctor assistants, physician assistants or other support personnel in the Department of Radiology that raise managing image acquisition related questions.
* Individuals that consent to participating in the study.
* Individuals scheduled to work at locations at Sending Extensions, Receiving Extensions and Control Extensions.

Exclusion Criteria:

* Individuals not able to understand or not willing to sign the informed consent form.
* Individuals that indicate that they do no comprehend RadConnect and/or its intended use after two educational sessions.
* Individuals not able to not willing to comply with the intended use of RadConnect.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are not patients, but radiologists, technologist, doctor assistants and physician assistants employeed by LUMC. That drive the radiological workflow and frequently raise and answer questions related to the image acquisition.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that adoption of RadConnect leads to reduction of phone calls to radiologists. | Numbers are continously measured during each shift of the subjects over a period of 40 consecutive working days during the before (phase 1) and 40 consecutive working days during the after phase (phase 2) of this study.
  * P1 = Mean number of calls per working day during regular working hours between Sending Extensions and Receiving Extensions in Before Phase
  * P2 = Mean number of calls per working day during regular working hours between Sending Extensions and Receiving Extensions in After Phase
  The primary endpoint will be obtained by testing the hypothesis that P1 > P2 using Wilcoxon's one-tailed test with significance level P < 0.05.

SECONDARY OUTCOMES:
Compare experiences and attitudes of technicians and radiologists towards RadConnect versus phone calls. | Continously measured during each shift of the subjects over a period of 40 consecutive working days during the before (phase 1) and 40 consecutive working days during the after phase(phase 2) of this study.
  * C1 = Mean number of calls per working day during regular working hours between Sending Extensions and Control Extensions in Before Phase
  * C2 = Mean number of calls per working day during regular working hours between Sending Extensions and Control Extensions in After Phase
  The first secondary endpoint will be obtained by testing the hypothesis that C1 ≠ C2 using Wilcoxon's two-tailed test with significance level P < 0.05.
Measure the characteristics of technician questions raised over phone and through RadConnect. | Continously measured during each shift of the subjects over a period of 40 consecutive working days during the before phase (phase 1) and 40 consecutive working days during the after phase (phase 2) of this study.
  • R2 = Mean number of completed RadConnect consultations per working day during regular working hours between Sending Extensions and Receiving Extensions in After Phase
  The second secondary endpoint will be obtained by testing the hypothesis that P1 ≠ P2 + R2 using Wilcoxon's two-tailed test with significance level P < 0.05.
Consolidated opinion usability and experience of RadConnect in itself and in comparison to alternative communication methods. | 1 hour, after completion of the after phase (phase 2 of this study)
  The third secondary endpoint will be obtained by aggregating survey responses. In the structured online survey, if more than half of the respondents indicate that they prefer communication over RadConnect to calling, it will be concluded that RadConnect is a viable alternative to calling. If more than half of radiologist respondents indicate that they believe RadConnect helps them avoid interruptions, it will be concluded that RadConnect is a viable alternative to calling that may help reduce radiologist interruptions. The opinions of study participants are captured as Likert scale response and averaged to obtain a consolidated opinion. The consolidated responses are visualized as histograms.

CONTACTS AND LOCATIONS:
Overall Officials: Hildo Lamb, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No